CLINICAL TRIAL: NCT04181892
Title: The Effects of Connective Tissue Graft Position on Clinical and Aesthetical Outcomes of Gingival Recession Treatment. A Controlled Randomized Clinical Trial
Brief Title: Effect of Connective Tissue Graft Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Mustafa Ozcan, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CukurovaU-PER-I
Record Dates: First submitted 2019-11-13; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Gingival Recession
Keywords: connective tissue graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+ CTG positioned apical to the CEJ (Experimental): Connective tissue graft covered by a coronally advanced flap which CTG apical of the CEJ level
  Interventions: Procedure: Coronally advanced flap + connective tissue graft
- CAF+CTG positioned on the CEJ (Other): Connective tissue graft covered by a coronally advanced flap which CTG on the CEJ level
  Interventions: Procedure: Coronally advanced flap + connective tissue graft

INTERVENTIONS:
Procedure: Coronally advanced flap + connective tissue graft — connective tissue graft covered by a coronally advanced flap with connective tissue graft apical of the cementoenamel junction level

SUMMARY:
Aim: The aim of this study was to compare the root coverage and aesthetic results of CAF+ CTG positioned apical to the CEJ (CAF+CTG-ACEJ) with CAF+CTG positioned on the CEJ (CAF+CTG-CEJ) for treating isolated gingival recession defects.

Methods: Thirthy-eight patients with Miller class I and II gingival recessions were enrolled. 19 patients were randomly assigned to the CAF+CTG-ACEJ group or CAF+CTG-CEJ group. Clinical and aesthetical evaluations were made at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age,

  * Periodontally and systemically healthy,
  * FMPS and FMBS <15%,
  * Presence of Miller Class I/II GR defect (≥3 mm in depth) at the buccal aspect of incisors and canines,
  * Presence of identifiable CEJ (step ≤1 mm at CEJ level and/or presence of a root irregularity/abrasion with identifiable CEJ, was accepted),
  * No previous periodontal surgery.

Exclusion Criteria:

* Smoking,
* Contraindications for surgery,
* Presence of recession defects associated with caries, deep abrasion, restoration or pulpal pathology.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Gingival Recession depth in millimeters | 6 months
  measured from the cemento-enamel junction to the gingival margin
keratinized tissue height in millimeters | 6 months
  measured from the mucogingival junction to the gingival margin
aesthetic evaluation assesed by visual analog scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ucak Turer, PhD, Principal Investigator — Professor
Locations (1):
- Cukurova University Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No